CLINICAL TRIAL: NCT00088075
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of the Efficacy and Safety of Risperidone for the Treatment of Schizophrenia in Adolescents
Brief Title: Investigate Risperidone for the Treatment of Schizophrenia in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003370
Record Dates: First submitted 2004-07-19; First posted 2004-07-21 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Adolescents
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
A clinical study to evaluate the efficacy, safety and tolerability of two dose ranges of risperidone (1 to 3 mg/day, and 4 to 6 mg/day) versus placebo (an inactive substance like a sugar pill) in adolescents (aged 13 to 17 years) with schizophrenia (i.e. abnormal behavior and thoughts). The study duration is about 6 to 7 weeks.

DETAILED DESCRIPTION:
Subjects will be aged 13 to 17 years with a diagnosis of schizophrenia. On enrollment, subjects will be assigned to receive 1 of 3 treatments (oral placebo tablets, oral risperidone tablets 1 to 3 mg, or oral risperidone tablets 4 to 6 mg), which will be administered daily for 6 weeks. Study medication will be increased to within the target dosage range during the first 7 days and then further increased until the maximum tolerated dose is achieved by day 14. The maximum tolerated dose will be maintained for the last 4 weeks of the study, unless dose adjustments are agreed with the Sponsor. Risperidone (1 to 3 mg or 4 to 6 mg) or placebo given orally as 0.5, 1, 2, 3, or 4 ,g tablets (or matching placebo) each day for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* A responsible person must be available to accompany the subject to the site at each visit
* patient must meet the DSM-IV criteria for schizophrenia

Exclusion Criteria:

* Patients with mild, moderate or severe mental retardation
* patients with a known or suspected history of substance dependence
* subjects weighing <35kg
* subjects who cannot swallow oral tablets

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2004-08; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in total PANSS (Positive and Negative Syndrome Scale for Schizophrenia) from baseline to the 6-week endpoint

SECONDARY OUTCOMES:
Change from baseline in PANSS subscale scores and Clinical Global Impression (CGI-S and CGI-I) scores, number of subjects achieving a clinical response (at least 20% improvement in total PANSS), safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Haas M, Unis AS, Armenteros J, Copenhaver MD, Quiroz JA, Kushner SF. A 6-week, randomized, double-blind, placebo-controlled study of the efficacy and safety of risperidone in adolescents with schizophrenia. J Child Adolesc Psychopharmacol. 2009 Dec;19(6):611-21. doi: 10.1089/cap.2008.0144. PMID 20035579
- See also: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of the Efficacy and Safety of Risperidone for the Treatment of Schizophrenia in Adolescents — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=523&filename=CR003370_CSR.pdf